CLINICAL TRIAL: NCT03644537
Title: Correlation Between Root Resorption and Dentin Sialoprotein Upon Application of Different Orthodontic Forces, a Split-mouth Technique, a Randomized Clinical Trial
Brief Title: Correlation Between Root Resorption and Dentin Sialoprotein Upon Application of Different Orthodontic Forces.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aya Ahmed Moursi El Faham (Other)
Responsible Party: Sponsor-Investigator, Aya Ahmed Moursi El Faham, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-07-13
Record Dates: First submitted 2018-07-13; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Root Resorption
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- heavy force 100gm (Other): heavy intrusive force is to be applied on a first premolar on one side
  Interventions: Procedure: Orthodontic intrusion
- medium force 25 gm (Other): medium intrusive force is to be applied on a first premolar on one side
  Interventions: Procedure: Orthodontic intrusion
- light force 10 gm (Other): light intrusive force is to be applied on a first premolar on one side
  Interventions: Procedure: Orthodontic intrusion

INTERVENTIONS:
Procedure: Orthodontic intrusion — 27 female patients coming to the Orthodontic department, Cairo University seeking orthodontic treatment, where their age ranges from 15 - 18 years, where their treatment plan include extraction of upper first premolars, and using the split-mouth technique, one side will be control group without application of force where the other side will receive intrusive mechanics for the same patient in the upper arch (one side will not receive any force and the same tooth on the other side of the arch will suffer intrusive mechanics, that's why named SPLIT MOUTH TECHNIQUE - as if the arch is split into two subjects, one control subject (tooth) and the other study subject (tooth) . According to the amount of force of the working side, the total number of patients will be divided into 3 groups.
  Each of 9 subjects, the first group where a light force will be applied (10 gm), the second group where moderate force will be applied (25gm), the third group where heavy force will be applied(100 gram).

SUMMARY:
Since root resorption is a frequent consequence of orthodontic treatment, DSP are non-collagenous dentin-specific matrix proteins postulated to be involved in the mineralization of pre-dentin into dentin. Calculating the amount of DSP -Dentine Sialo Protein- produced upon root resorption might be an indicative biological marker for root resorption

DETAILED DESCRIPTION:
Histological and radiographic observations have shown that root resorption is a frequent consequence of orthodontic treatment (Reitan, 1974; Rygh, 1977; Harry and Sims, 1982). In most patients this resorption is minor and of no importance. A few teeth however exhibit severe resorption. In a study by Goldson and Henrikson (1975) it was found that 6 per cent of 924 teeth were resorped more than 2 mm after treatment with a Begg appliance and Malmgren et al. ( 1982) found a similar degree of root resorption in 10 percent of 264 incisors treated with an edgewise appliance and in 5 percent of 176 incisors treated with a Begg appliance(1).

Root resorption resulting from undesirable orthodontic force is an unwanted sequele , that fears all orthodontists including their experts as well(2).

DSP are non-collagenous dentin-specific matrix proteins postulated to be involved in the mineralization of pre-dentin into dentin (3,4) .Dentin undergoes continuous deposition throughout life as a secondary dentin only on the pulpal surface. Therefore, these proteins are not routinely released into the surrounding space as dentin does not undergo the process of remodeling as in bone. It is only in the presence of active external root resorption that these proteins could be freed into the periodontal ligament space(5).

Since periapical -intraoral- radiograph gives a two dimensional information, which detect root resorption after 60- 70% of the mineralized tissue is lost. (6) So, it's not sensitive in detecting early root resorption so in this study the investigators introduce the biological marker DSP to monitor root resorption from its onset by collecting samples from the GCF -gingival crevicular fluid- for its detection.

Calculating the amount of DSP -Dentine Sialo Protein- produced upon root resorption might be an indicative biological marker for root resorption.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent female patients age ranging from 15- 18 yrs, with the full set of the permanent dentition.
* No previous orthodontic treatment.
* Class I crowding or Class II malocclusion whose treatment requires extraction of first maxillary premolars.
* Adequate oral hygiene.

Exclusion Criteria:

* Systematic diseases.
* Bad Oral hygiene.
* Missing permanent teeth (except for third molars).
* Uncontrolled Pathological Conditions that may contra-indicate immediate orthodontic treatment (caries, gingivitis, periodontitis).

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-10-07 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
DSP (DentinSialoProtein ) | with in 3 monthes from applied intrusion
  concentration of DSP is expected to be secreted into the gingival crevicular fluid upon root resorption

CONTACTS AND LOCATIONS:
Locations (1):
- economic treatment center, Orthodontics Department, Cairo University, Cairo, Egypt